CLINICAL TRIAL: NCT01587027
Title: The Safety Evaluation of Aminophylline and Methazolamide When Administered Orally Alone and in Combination to Healthy Volunteers
Brief Title: Safety Evaluation of Aminophylline and Methazolamide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poudre Valley Health System (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Gary J. Luckasen, MD, Prinicipal Investigator, Poudre Valley Health System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GQ01 DARPA
Record Dates: First submitted 2012-04-16; First posted 2012-04-27 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Mountain Sickness
Keywords: Altitude Sickness; High Altitude Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Aminophylline; Theophylline; Methazolamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence A (Active Comparator): Aminophylline, Methazolamide, Aminophylline and Methazolamide
  Interventions: Drug: Aminophylline; Drug: Methazolamide; Drug: Aminophylline and Methazolamide
- Sequence B (Active Comparator): Methazolamide, Aminophylline, Aminophylline and Mathazolamide
  Interventions: Drug: Aminophylline; Drug: Methazolamide; Drug: Aminophylline and Methazolamide

INTERVENTIONS:
Drug: Aminophylline — Aminophylline dosage form-tablet dosage-500mg
  Other Names: theophylline
Drug: Methazolamide — Methazolamide dosage form-tablet dosage-250mg
  Other Names: Neptazane
Drug: Aminophylline and Methazolamide — Aminophylline 500mg orally and Methazolamide 250mg orally
  Other Names: theophylline; Neptazane

SUMMARY:
This safety study is the first in a series of studies testing the application of the combination of aminophylline and methazolamide.

DETAILED DESCRIPTION:
After successful completion of this safety trial, our goal will be to evaluate the safety of this combination in healthy individuals exposed to hypoxia and exercise. Subsequently, an efficacy study will clarify whether this drug combination improves physical and mental functions in human subjects under high altitude conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be healthy non-smoking adult male and female volunteers between the ages of 18 and 40 years, with a BMI of 18-30 kg/m2 and weighting at least 150 lbs. Women who are of childbearing potential, must, if sexually active, must agree to use appropriate contraceptive measures for the duration of the study and for one (1) month afterwards.
* Subjects must agree not to donate blood, plasma, platelets, or any other blood components during the study and for 4 weeks after the last dose.

Exclusion Criteria:

* History or manifestation of clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematologic or other medical disorders.
* Serious mental or physical illness within the past year.
* History of clinically significant illness within 4 weeks prior to Day 1.
* History of allergic reaction, hypersensitivity or idiosyncratic reaction to any of the products administered during the study, including allergy to any sulfa or sulfonamide derivatives.
* Use of any of the following:
* Any concomitant medication. Subjects who have received any prescribed or non-prescribed (over-the-counter [OTC]) systemic medication, topical medications, or herbal supplements within 14 days from Day 1. St. John's Wort (hypericin) must not have been taken for at least 30 days prior to Period 1, Day 1.
* Any drugs, foods or substances known to be strong inhibitors or strong inducers of CYP enzymes (also known as cytochrome P450 enzymes); especially CYP 1A2, or Pgp within 30 days prior to Period 1, Day 1.
* Currently abusing drugs or alcohol or with a history of drug or alcohol abuse within the past two years.
* Positive results on screening tests for drugs of abuse, cotinine or alcohol at screening or the pre-dose assessment at check-in.
* Clinically significant ECG abnormality, in the opinion of the Investigator.
* Use of tobacco products or other nicotine-containing products (including smoking cessation aids, such as gums or patches) with in 14 days of screening and throughout hospitalization.
* Subjects of childbearing potential who are pregnant (as based on test results) or are breast feeding.
* Has taken any other investigational drug during the 30 days prior to the screening visit or is currently participating in another investigational clinical trial.
* Subjects who have made any significant donation (including plasma) or have had a significant loss of blood within 30 days prior to Period 1, Day 1.

Receipt of a transfusion or any blood products within 30 days prior to Period 1, Day 1.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Luckasen, M.D., Principal Investigator — Poudre Valley Health System
Locations (1):
- Medical Center of the Rockies, Loveland, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://pvhs.org/research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study proposed to randomize approximately 24 subjects to complete 16.
Pre-assignment Details: A total of 26 subjects were screened and consented. Of the subjects assessed, 21 (81%) passed and 5 (19%) were screen failures. Of those subjects who were screen failures, 3 (60%) had abnormal lab results and 2 (40%) had scheduling difficulties.
Groups:
- Sequence A: Treatment 1, Treatment 2, Treatment 3
  Treatment 1 : Aminophylline dosage form-tablet dosage-500mg
  Treatment 3 : Aminophylline 500mg orally and Methazolamide 250mg orally
- Sequence B: Treatment 2, Treatment 1, Treatment 3
  Treatment 3 : Aminophylline 500mg orally and Methazolamide 250mg orally
  Treatment 2 : Methazolamide dosage form-tablet dosage-250mg
Period: First Intervention (1 Day)
Arm/Group | Sequence A | Sequence B
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout (1 Day)
Arm/Group | Sequence A | Sequence B
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Sequence A | Sequence B
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Washout (1 Day)
Arm/Group | Sequence A | Sequence B
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Sequence A | Sequence B
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Discharge (1 Day)
Arm/Group | Sequence A | Sequence B
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants must be healthy non-smoking adult male and female volunteers between the ages of 18 and 40 years, with a BMI of 18-30 kg/m2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants] — Age=between 18 and 40.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 8 | 8 | 16
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.60429 (5.12602) | 25 (3.16228) | 25.125 (3.96443)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
BMI = <=18-30 kg/m2 [Number; unit: Participants] | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events.
Description: Adverse event data was evaluated for incidence and severity for 6 days.
Time Frame: 6 days.
Population: All enrolled participants were analyzed for adverse events.
Measure: Number; unit: Events
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 8 | 8
Events | 29 | 40

ADVERSE EVENTS:
Time Frame: 6 days per subject.
Description: Participants were monitored for adverse events during 6 days of study participation.
Groups:
- Arm A: Aminophylline (1 Day) Washout (1 Day) Methazolamide (1 Day) Washout (1 Day) Both Aminophylline & Methazolamide (1 Day) Discharge (1 Day)
- Arm B: Methazolamide (1 Day) Washout (1 Day) Aminophylline (1 Day) Washout (1 Day) Both Aminophylline & Methazolamide (1 Day) Discharge (1 Day)
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=8) | Arm B (N=8)
Blister at IV site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decreased visual acuity (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness when standing (Nervous system disorders) | 1 (1) | 0 (0)
Drunk feeling (Nervous system disorders) | 0 (0) | 1 (1)
Facial tingling (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (6) | 5 (10)
Jitteriness (Nervous system disorders) | 4 (6) | 7 (9)
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Numbness (Nervous system disorders) | 2 (2) | 1 (1)
Pain & edema to venipuncture site (Nervous system disorders) | 1 (1) | 0 (0)
Pain at IV site (Nervous system disorders) | 1 (1) | 0 (0)
Pressure in forearms (Nervous system disorders) | 0 (0) | 1 (1)
Shoulder stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 3 (3) | 4 (7)
Lightheadedness (Nervous system disorders) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No